CLINICAL TRIAL: NCT01522846
Title: Influence by Heparinized Flush Solution of the Radial Artery Catheter: INTEM and HEPTEM Analysis.
Brief Title: Heparin Solution and INTEM/HEPTEM Analysis
Status: Completed | Type: Observational
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Hyo-Seok Na, Assistant professor, Seoul National University Bundang Hospital
Other Study IDs: B_1112_069_003
Record Dates: First submitted 2012-01-09; First posted 2012-02-01 (Estimated); Last update posted 2013-08-29 (Estimated); Status verified 2013-08

CONDITIONS: Brain Tumor; Spinal Stenosis; Cerebral Artery Anuerysm
MeSH Terms: conditions — Brain Neoplasms; Spinal Stenosis | interventions — Heparin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Heparin
  Interventions: Drug: Heparin

INTERVENTIONS:
Drug: Heparin — Heparinized flush solution contained heparin concentration of 2 unit/ml and continuous flow of the flush solution was 5 ml/h at 300 mmHg.

SUMMARY:
Heparinized solution has been used for maintenance of arterial catheter during perioperative period. Although the infused dose of heparin is very low, the investigators examine whether the heparin effect is remained or not in blood using rotational thromboelastometry (ROTEM) analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring continuous invasive arterial pressure monitoring during operation for anesthetic management.

Exclusion Criteria:

* heparin hypersensitivity
* hematologic disease
* anticoagulant medication

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients requiring continuous invasive arterial pressure monitoring during operation for anesthetic management.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2012-01; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
INTEM test | at 30 min before operation and 30 min after operation
  INTEM is not an abbriviation. INTEM is one of the ROTEM test and it is an coagulation test name (such as prothrombin time test) using patient's whole blood. We put the blood sample of patinet into the machine, so the result comes out automatically. It will be checked twice at pre- and postopertive 30 minute and it'll be analyzed and compared.
HEPTEM test | at 30 min before operation and 30 min after operation
  HEPTEM is not an abbriviation. HEPTEM is one of the ROTEM test and it is an coagulation test name (such as prothrombin time test) using patient's whole blood. We put the blood sample of patinet into the machine, so the result comes out automatically. It will be checked twice at pre- and postopertive 30 minute and it'll be analyzed and compared.

SECONDARY OUTCOMES:
Total infused units of heparin | periond from starting operation to finishing operation (espected average of 5 hours).

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seonnam, Gyounggi, South Korea